CLINICAL TRIAL: NCT02321332
Title: Unilateral Sequential Versus Bilateral Simultaneous Sympathectomy for Palmar Hyperhidrosis: a Study of 407 Cases.
Brief Title: Unilateral Sequential Sympathectomy for Palmar Hyperhidrosis
Acronym: ETS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tmaer Youssef Mohamed (Other)
Responsible Party: Sponsor-Investigator, Tmaer Youssef Mohamed, assistant professor of surgery, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MFM2010344
Record Dates: First submitted 2014-12-11; First posted 2014-12-22 (Estimated); Last update posted 2014-12-22 (Estimated); Status verified 2014-12

CONDITIONS: Palmar Hyperhidrosis
Keywords: Palmar hyperhidrosis; Endoscopic thoracic sympathectomy

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- B-ETS (Active Comparator): Bilateral simultaneous endoscopic thoracic sympathectomy: bilateral simultaneous T2-T3 ganglionectomy.
  Interventions: Procedure: bilateral simultaneous endoscopic thoracic symapthectomy
- S-ETS (Active Comparator): unilateral sequential endoscopic thoracic sympathectomy: unilateral T2-T3 ganglionectomy of the dominant side followed by T2-T3 ganglionectomy of the other side after 2 months interval
  Interventions: Procedure: unilateral sequential endoscopic thoracic symapthectomy.

INTERVENTIONS:
Procedure: bilateral simultaneous endoscopic thoracic symapthectomy — Patients underwent bilateral simultaneous T2-T3 ganglionectomy using thoracoscopic approach.
  Arms: B-ETS
Procedure: unilateral sequential endoscopic thoracic symapthectomy. — Patients underwent unilateral T2-T3 ganglionectomy of the dominant side followed by T2-T3 ganglionectomy of the other side after 2 months interval.
  Arms: S-ETS

SUMMARY:
Comparison between unilateral sequential and bilateral simultaneous endoscopic thoracic sympathectomy for palmar hyperhidrosis on patients outcomes notably compensatory hyperhidrosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering palmar hyperhidrosis

Exclusion Criteria:

* Patients with pleural adhesions, bleeding diathesis, local infection or previous operation for hyperhidrosis

Ages: 8 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Actual)
Dates: Start 2010-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Number of participants developing compensatory hyperhidrosis (reflex sweating) following sympathectomy. | one year
  Number pf patients developing compensatory hyperhidrosis (reflex sweating) following sympathectomy. Compensatory hyperhidrosis was graded as "severe" when the patient mentioned that sweating interfered with his or her normal activity, "moderate" when the patient indicated that his or her sweating was not bothersome and "mild" when the patient did not mention dampness or made only a brief reference.

SECONDARY OUTCOMES:
Number of patients who will be satisfied or unsatisfied regarding the procedure. | one year
  we measure patient satisfaction regarding the procedure by asking the patients to rate their level of satisfaction as very satisfied, somewhat satisfied, somewhat dissatisfied and very dissatisfied. Patients were considered satisfied if they reported being very satisfied or somewhat satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: tamer youssef, MD, Study Director — Mansoura Faculty of Medicine